CLINICAL TRIAL: NCT03890198
Title: A Phase 1, Open-Label Study Evaluating the Safety, Tolerability and Efficacy of LCAR-C182A, an Anti-Claudin18.2 CAR-T Cell Therapy in Patients With Advanced Gastric Cancer and Pancreatic Ductal Adenocarcinoma
Brief Title: A Phase 1 Study of LCAR-C182A Cells in the Treatment of Advanced Gastric Cancer and Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: the Preliminary data, progress of this study and the adjustment of the pipeline and strategy .
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO-GPC01
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Gastric Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Gastric cancer; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chimeric Antigen Receptor T cell (Experimental): LCAR-C182A Cells
  Interventions: Biological: LCAR-C182A cells

INTERVENTIONS:
Biological: LCAR-C182A cells — Patients receive fludarabine (3×300 mg/ m^2) and cyclophosphamide (3×30 mg/m^2) IV on days -5 to-3, and then Patients receive CAR-T cells. PS：The specific dose of fludarabine and cyclophosphamide is adjusted according to the individual condition of the subject and the judgment of the investigator.

SUMMARY:
This is an open label, single center, single arm phase 1 study to evaluate the safety , tolerability, pharmacokinetics and efficacy and immunogenicity of LCAR-C182A cells targeting Claudin18.2 in the treatment of patients with advanced gastric cancer and Pancreatic Ductal Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. the subject has fully understood the possible risks and benefits of participating in this study, and has signed informed consent form (ICF);
2. Age 18-75 years;
3. Histologically confirmed unresectable advanced gastric adenocarcinoma (including gastric esophageal junction adenocarcinoma) or advanced pancreatic ductal carcinoma;
4. Claudin18.2 positive by immunohistochemistry;
5. Previously accepted the recommendations of the national comprehensive cancer network (NCCN 2019 V1) or the gastric cancer guidelines of the cooperative professional committee on clinical oncology (CSCO 2018 V1) of the Chinese anti-cancer association, or the standard treatment regimen considered to be equivalent by the investigator；
6. Pancreatic cancer: ≥1 line standard chemotherapy, or regimens considered equivalent by the investigator, have recently failed or cannot be tolerated in the first line；
7. By CT scan or MRI, patients with a measurable lesion ≥1cm or a single lymph node with a short diameter ≥1.5cm (RECIST 1.1) are required to obtain permission from the principal investigator if the lesion is measurable, i.e. the target lesion is lymph node metastasis；
8. ECOG 0 ~ 1;
9. expected survival period≥ 3 months；
10. blood routine was in line with the certain standards；
11. blood biochemical test meets the certain criteria；
12. blood pregnancy test of women of child-bearing age was negative；

Exclusion Criteria:

1. has received CAR-T therapy targeting any target.
2. ever received any treatment targeting Claudin18.2.
3. brain metastasis with central nervous system symptoms;
4. pregnant or lactating women;
5. uncontrolled diabetes;
6. Oxygen absorption is required to maintain adequate blood oxygen saturation;
7. Patients with pyloric obstruction, gastric perforation, partial or complete intestinal obstruction and complete biliary obstruction that cannot be relieved after active treatment;
8. Hepatic disease;Chronic hepatitis infection with HBV/HCV;
9. Seropositive for human immunodeficiency virus (HIV);
10. Any active autoimmune disease or history of autoimmune disease;
11. have obvious bleeding tendency, such as gastrointestinal bleeding, coagulation dysfunction, and hypersplenism;
12. unstable angina within the past 6 months, symptomatic congestive heart failure or myocardial infarction;
13. severe uncontrolled arrhythmias;Left ventricular ejection fraction <50%;
14. activity requiring parenteral antibiotics or uncontrolled infection;There is evidence of severe active viral, bacterial or uncontrolled systemic fungal infection
15. other malignancies in the past 5 years except for non-melanoma skin cancer or in-situ cervical cancer;
16. chronic diseases treated with steroids or other immunosuppressive agents;
17. Concurrent use of hematopoietic growth factor;
18. Concurrent use of anticancer drugs or therapy (except radiotherapy for pain relief, etc., for non-target lesions);
19. Concurrent investigational treatment;
20. Have undergone chemotherapy, radiotherapy, or other experimental treatment within 4 weeks prior to apheresis
21. stroke or convulsion within 6 months before signing ICF;
22. Have received any live, attenuated vaccine within 4 weeks prior to apheresis;
23. Have underwent major surgical operation within 2 weeks prior to apheresis, or anticipate to undergo a major surgical operation during the study process or within 2 weeks posterior to study treatment (with the exception of anticipated local anesthesia surgery)
24. Allergic to the study drug expient and related expients (including but not limited to DMSO and dextran 40), or allergic to other immunotherapy and related drugs
25. Presence of any condition that, in the opinion of the investigator, would prohibit the patient from undergoing treatment under this protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 90 days post infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product,and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
MTD）/ RP2D regimen finding | 90 days post infusion
  Maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D)
Transgene Levels of LCAR-C182A CAR-T Cells | 2 years post infusion
  Transgene Levels of LCAR-C182A CAR-T Cells using sensitive assay methods will be assessed
Chimeric Antigen Receptor T (CAR-T) Positive Cell Concentration | 2 years post infusion
  Venous blood samples will be collected for measurement of CAR-T positive cellular concentration
Systemic Cytokine Concentrations | 2 years post infusion
  Serum cytokine concentrations such as IL-2, IL-6, IL-8, 1L-10, TNF-α, IFN-γ will be measured for biomarker assessment

SECONDARY OUTCOMES:
Overall response rate (ORR) after administration | 2 years post infusion
  The ORR is defined as the proportion of patients with complete or partial response according to Response Evaluation Criteria In Solid Tumors（RECIST) criteria.
Duration of remission (DOR) after administration | 2 years post infusion
  The DOR is defined as the time between the initial onset of complete or partial remission and the onset of disease progression in patients with objective remission according to Response Evaluation Criteria In Solid Tumors（RECIST) criteria.
Progress Free Survival (PFS) after administration | 2 years post infusion
  The PFS is defined as the Time from enrollment until disease progression or death according to Response Evaluation Criteria In Solid Tumors（RECIST) criteria.
Overall Survival (OS) after administration | 2 years post infusion
  The OS is defined as Time from enrollment until death from any cause according to Response Evaluation Criteria In Solid Tumors（RECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Enxiao Li, MD,PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi, China